CLINICAL TRIAL: NCT00129753
Title: Phase II Study of Alemtuzumab (Campath-1H) Monoclonal Antibody in Patients With Relapsed and Resistant Classical Hodgkin's Disease
Brief Title: Alemtuzumab (Campath-1H) Monoclonal Antibody in Patients With Relapsed and Resistant Classical Hodgkin's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Anas Younes, M.D. / Professor, UT MD Anderson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0742
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Hodgkin's Disease; Lymphoma
Keywords: Campath-1H Monoclonal Antibody; Alemtuzumab; Campath; Campath-1H; Relapsed and Resistant Classical Hodgkin's Disease; Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma; Recurrence | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alemtuzumab (Experimental)
  Interventions: Drug: Alemtuzumab (Campath-1H)

INTERVENTIONS:
Drug: Alemtuzumab (Campath-1H) — Escalating dose 3mg, 10 mg, 30 mg on three consecutive days, then 30 mg three times per week by subcutaneous injections for 12 weeks. Each 30 mg dose will be divided in 2 injections to be administered in each thigh.
  Other Names: Campath; Campath-1H; Campath-1H Monoclonal Antibody

SUMMARY:
Primary Objective:

To determine the safety and efficacy of Campath-1H (Alemtuzumab) in patients with relapsed and resistant classical Hodgkin's lymphoma.

Secondary Objectives:

1. To determine the duration of response and time to progression after Campath-1H therapy in this patient population.
2. To determine the effect of Campath-1H on serum IL-6, IL-10, and IL-13 levels in patients with relapsed and resistant classical Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Alemtuzumab is the type of drug known as a "monoclonal antibody". The antibody binds to a specific protein (antigen) called CD52. CD52 is found on the surface of normal lymphocytes and monocytes. When the antibody binds to the protein on the surface of the lymphocyte or monocyte it causes the cell to die. The goal of the study is to learn if killing normal lymphocytes and monocytes with alemtuzumab will result in regression (lessening) of the cancer cells.

Alemtuzumab is usually given by an infusion into a vein. However, in this study, it will be given as an injection under-the-skin. This method of giving alemtuzumab is not approved by the FDA. The purpose of giving the drug by injection under the skin is to decrease the side effects observed with infusion by vein.

Before you can start treatment on this study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical exam Blood (about 2 tablespoons) will be collected for routine tests. A bone marrow sample will be collected to learn if your Hodgkin's lymphoma has spread to the bone marrow. To collect a bone marrow sample (biopsy), an area of the hip bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. A CT scan or MRI of the chest, abdomen (stomach), and pelvis (waist area) will be done. You will also have a PET scan or a Gallium scan to check on the status of the disease. You will be required to have a heart scan or an echocardiogram to check how strong your heart muscle is. You will be asked about medications that you are currently taking, including over-the-counter medications. Women who are able to have children must have a negative blood pregnancy test.

If you are found to be eligible to take part in this study, you will receive alemtuzumab 3 times a week as an injection under the skin. Typically these injections will be given on Monday, Wednesday, and Friday. Each dose will be divided into two injections to be given in each thigh. You will be treated for 12 weeks in a row. The treatment doses will be given by a nurse at M. D. Anderson in an outpatient setting. Before each injection, you may receive Tylenol and/or Benadryl to decrease the risk of side effects caused by the study drug.

During the 12-week treatment course, in addition to your study drug injections, you will visit the clinic every 3 weeks for physical exam and routine blood tests (2 tablespoons each). You will also have a blood test (1 tablespoonful) every week to find out if you are having a certain type of viral infection (cytomegalovirus, called CMV). If your blood tests show that your CMV blood levels are increasing, you may need treatment with anti-viral antibiotics to control your viral infection. You doctor will also give you antibiotics to take by mouth to prevent possible infections.

If the tumor grows during treatment or you experience any intolerable (very bad) side effects, you will be taken off study and your doctor will discuss other treatment options with you.

Within 3 weeks of the last dose of alemtuzumab, you will have a physical exam, routine blood tests (2 tablespoons), CT scans of the chest, abdomen, and pelvis, and a bone marrow biopsy (if needed). These tests will help show whether your tumor is shrinking after therapy. If these tests show that your tumor is not growing, you will be placed on observation and your tumor status will be checked up on every 3 months by repeating similar tests.

This is an investigational study. Alemtuzumab is FDA approved for the treatment of chronic lymphocytic leukemia and is commercially available. However, the FDA has not approved alemtuzumab for the treatment of Hodgkin's disease. Furthermore, the FDA has not approved the injection of alemtuzumab under the skin for the treatment of cancer. A maximum of 35 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory Hodgkin's disease with a minimum of 2 prior treatment regimens, including autologous bone marrow transplantation.
* Must have histologically proven diagnosis of nodular sclerosis or mixed cellularity Hodgkin's disease.
* Hodgkin's lymphoma should be limited to lymph nodes, spleen, and bone marrow.
* Must have bi-dimensionally measurable disease defined as a lymph node at least 2 cm by computed tomography (CT) scan.
* Platelet count equal to or greater than 50,000/uL; absolute neutrophil count equal to or greater than 1,000/uL.
* Must sign a consent form.
* Males or females equal to or greater than 18 years of age.
* Patients may be taking voriconazole, itraconazole, or diflucan.

Exclusion Criteria:

* No serious inter-current infections requiring therapy.
* No Hodgkin-specific therapy within the last 3 weeks.
* Pregnant women and women of childbearing potential and men of reproductive potential who are not practicing adequate contraception.
* Lymphocyte depletion or lymphocyte predominance histology.
* History of HIV infection.
* Central nervous system (CNS) involvement with lymphoma including epidural disease and cord compression.
* Prior allogeneic stem cell transplantation.
* Patients receiving steroids within 3 weeks of registration.
* Patients with a history of prior severe opportunistic infections that are controlled by T-cell immunity, such as pneumocystis pneumonia (PCP), herpes virus infections, mycobacterial disease, invasive mold infections or endemic fungi.
* Patients with an ejection fraction of less than 40%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-06-22 (Actual); Primary Completion 2006-09-05 (Actual); Study Completion 2006-09-05 (Actual)

PRIMARY OUTCOMES:
Response Rate | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Anas Younes, M.D., Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org